CLINICAL TRIAL: NCT03568383
Title: Protecting Households On Exposure to Newly Diagnosed Index Multidrug-Resistant Tuberculosis Patients (PHOENIx MDR-TB)
Brief Title: Protecting Households On Exposure to Newly Diagnosed Index Multidrug-Resistant Tuberculosis Patients
Acronym: PHOENIx MDR-TB
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A5300B/I2003B/PHOENIx; 12041 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis, MDR
Keywords: Tuberculosis; Multidrug Resistance; Prevention; Household Contact
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis | interventions — OPC-67683; Isoniazid; Pyridoxine; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Delamanid (DLM) (Experimental): HHCs will receive delamanid (DLM) for 26 weeks.
  Interventions: Drug: Delamanid (DLM)
- Arm B: Isoniazid (INH) (Experimental): HHCs will receive isoniazid (INH) and pyridoxine (vitamin B6) for 26 weeks.
  Interventions: Drug: Isoniazid (INH); Dietary Supplement: Pyridoxine (vitamin B6)

INTERVENTIONS:
Drug: Delamanid (DLM) — Adults and children ≥30 kg: delamanid 200 mg orally once daily.
  Children ≥2.5 kg to <30 kg: weight-band dosing orally once daily as per the study protocol. As children gain weight, their DLM dose should be adjusted, typically every month or as the visit schedule permits.
  Arms: Arm A: Delamanid (DLM)
Drug: Isoniazid (INH) — Adults and children ≥24 kg: INH 300 mg orally once daily.
  Children ≥2.5 kg to <24 kg: INH weight-band dosing orally once daily as per the study protocol. As children gain weight, their INH dose should be adjusted.
  Arms: Arm B: Isoniazid (INH)
Dietary Supplement: Pyridoxine (vitamin B6) — All HHCs in Arm B must receive pyridoxine (vitamin B6) with each dose of INH based on the current local dosing guidelines. For children up to 3 years of age and nursing women, pyridoxine will be given as per local standard of care. Pyridoxine is not supplied through the study.
  Arms: Arm B: Isoniazid (INH)

SUMMARY:
The purpose of this study is to compare the efficacy and safety of 26 weeks of delamanid (DLM) versus 26 weeks of isoniazid (INH) for preventing confirmed or probable active tuberculosis (TB) during 96 weeks of follow-up among high-risk household contacts (HHCs) of adults with multidrug-resistant tuberculosis (MDR-TB) (index cases). High-risk HHCs are those with HIV or non-HIV immunosuppression, latent TB infection, and young children below the age of 5 years.

DETAILED DESCRIPTION:
This study will compare the efficacy and safety of 26 weeks of delamanid (DLM) versus 26 weeks of isoniazid (INH) for preventing confirmed or probable active tuberculosis (TB) during 96 weeks of follow-up among high-risk household contacts (HHCs) of adults with multidrug-resistant tuberculosis (MDR-TB) (index cases). High-risk HHCs are those with HIV or non-HIV immunosuppression, latent TB infection, and young children below the age of 5 years.

If at least one HHC within a household (HH) is found to be eligible, the HH will be randomized to one of the following:

Arm A: DLM daily for adults, adolescents, and children, given for 26 weeks.

Arm B: INH daily for adults, adolescents, and children, given for 26 weeks AND pyridoxine (vitamin B6) daily for adults, adolescents, and children, given for 26 weeks.

All high-risk HHCs in the same HH will receive the same randomized regimen.

All participants will be in the study for 96 weeks. At study entry, index cases will undergo a medical history review and sputum collection. HHCs will have study visits at study entry and at Weeks 2, 4, 8, 12, 16, 20, 26, 36, 48, 60, 72, 84, and 96. Visits may include physical examinations; blood, urine, and sputum collection; electrocardiograms (ECGs); and questionnaires and assessments. Forty HHCs under the age of 5 taking DLM will undergo an intensive PK visit at Week 8.

ELIGIBILITY:
Inclusion Criteria:

INDEX CASE

* Men and women age greater than or equal to 18 years.
* Pulmonary MDR-TB defined as:

  * Confirmation of rifampin/rifampicin (RIF) resistance and INH resistance by
  * adequate source documentation (including date of testing, test methodology, and test results) of RIF and INH resistance from a licensed/nationally approved* referral program, OR
  * if either or both results are unknown or not adequately documented (as noted above), then confirmation must be obtained using a DAIDS-approved laboratory that operates according to Good Clinical Laboratory Practices (GCLP) guidelines and participates in an appropriate external quality assurance (EQA) program.
  * *NOTE: The term "licensed/nationally approved" refers to a laboratory that has been certified or licensed by an oversight body within that country and approved for RIF and/or INH resistance testing.
  * NOTE: Pre-XDR and XDR TB are not exclusionary. See the A5300B/I2003B/PHOENIx MOPS for study-approved molecular and phenotypic methods.
* Started MDR-TB treatment within the past 90 days.
* Ability and willingness of the index case to provide informed consent to access the HH and approach HH members for evaluation.
* HH of index case has at least one reported HHC.

HOUSEHOLD CONTACTS

If any member(s) of the HH is/are not eligible or do not want to participate, all other eligible TB contacts within the HH can still participate.

* Currently lives or lived in the same dwelling unit or plot of land and shares or has shared the same housekeeping arrangements as the index case and who reports exposure within 90 days prior to the index case starting MDR-TB treatment. Also, shared greater than 4 hours of indoor airspace with the index case during any one-week period prior to the index case starting MDR-TB treatment.
* HHCs must be in one of the following high-risk groups:

  * All children 0 to less than 5 years old at the time of enrollment, regardless of LTBI or HIV status;
  * Adults, adolescents, and children greater than or equal to 5 years of age who are LTBI test positive (either TST-positive (greater than or equal to 5 mm) or IGRA-positive), and whose HIV status is negative, indeterminate, or unknown, and who are not non-HIV immunosuppressed;
  * NOTE: Both TST and IGRA testing are required for screening unless TST testing is not available due to global shortages or in-country supply challenges, but only one positive test is required for eligibility.
  * Adults, adolescents, and children greater than or equal to 5 years of age who are HIV-infected or are non-HIV immunosuppressed (defined as receiving anti-tumor necrosis factor (TNF) treatment, or being solid organ or hematologic transplant recipients), regardless of LTBI test status.
* HIV-1 infection status must be documented as positive, negative, indeterminate or unknown for all HHCs. Unknown status includes those who previously tested HIV negative but the test was performed more than one year ago. HIV testing will be offered to all HHCs with negative of unknown status. For adults (18 years and older), HIV-1 infection must be documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA viral load greater than 1000 copies/mL. Two or more plasma HIV-1 RNA viral loads of greater than 1,000 copies/mL are also acceptable as documentation of HIV infection. More information is available on this criterion in the protocol.
* The following specific laboratory values for infants, children, and adults obtained within 30 days prior to study entry by any DAIDS-approved non-US laboratory.

  * Absolute neutrophil count (ANC) greater than or equal to 750 cells/mm^3
  * Hemoglobin greater than or equal to 7.4 g/dL
  * Platelet count greater than or equal to 50,000/mm^3
  * Creatinine less than or equal to 2 × upper limit of normal (ULN)
  * Potassium level greater than or equal to 3.0 mEq/L
  * Aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) less than or equal to 3 × ULN
  * Total bilirubin less than or equal to 2.5 × ULN (Note: if on atazanavir (ATV), total bilirubin greater than 2.5 x ULN is permitted if direct bilirubin less than or equal to 2.5 × ULN)
  * Albumin greater than 3 g/dL
  * NOTE: Participants with results from other laboratory tests that are outside the normal range may be eligible for the study, at the discretion of the site investigator, if not considered to be an obstacle to entry.
* For females of reproductive potential, negative serum or urine pregnancy test within 7 days prior to study entry by any DAIDS-approved non-US laboratory that operates in accordance with GCLP and participates in appropriate external quality assurance programs.

  * NOTE: Reproductive potential is defined as:
  * Girls who have reached menarche or
  * Women who have had menses within the past 12 consecutive months and who do not have an FSH greater than 40 IU/L or
  * Women who have had menses within the past 24 consecutive months if an FSH measurement is not available
  * Women who have not undergone surgical sterilization (e.g., hysterectomy, or bilateral oophorectomy, or bilateral salpingectomy).
  * Female participants who are participating in sexual activity that could lead to pregnancy must agree to use one reliable form of contraceptive (i.e., hormonal contraceptive, condoms, IUD, diaphragm with spermicide, or cervical cap with spermicide) while receiving study treatments.
  * NOTE: Female participants who are not of reproductive potential, as defined above, or whose male partner(s) have undergone successful vasectomy with documented azoospermia or have documented azoospermia for any other reason, are eligible without requiring the use of contraceptives. Participant-reported history is acceptable documentation of menopause, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy.
* For infants (0 to 1 year of age), weight greater than or equal to 2.5 kg at screening.
* Ability and willingness of participant or legally-authorized representative (legal guardian or biological parent) to provide informed consent or assent as appropriate.
* Chest radiograph without evidence of active TB performed within 70 days prior to study entry for HHCs greater than or equal to 2 years of age and within 30 days prior to study entry for HHCs less than 2 years of age.
* QTcF interval less than or equal to 460 ms within 30 days prior to study entry as confirmed by the central ECG reading center.
* Enrollment of the HHC within 30 days after the index case is enrolled. In the event that a HHC is suspected of having TB, then this window for enrollment may be extended from within 30 days to within 70 days to allow for TB testing of the HHC.

Exclusion Criteria:

INDEX CASE

* Has previously enrolled into the A5300B/I2003B/PHOENIx trial as an index case or HHC, or is a member of a HH which has previously enrolled into the A5300B/I2003B/PHOENIx trial.

HOUSEHOLD CONTACTS

* Current confirmed or probable or possible pulmonary or extrapulmonary TB, based on the following criteria: the current ACTG Diagnosis Appendix 100 for adults and for children of greater than or equal to 15 years of age; or the modified pediatric TB definitions for children less than 15 years of age as described in the A5300B/I2003B/PHOENIx MOPS.
* Receipt of more than 30 cumulative days of INH, rifamycin, fluoroquinolone, or DLM in the 90 days prior to study entry.
* History of or current liver cirrhosis at any time prior to study entry.
* Evidence of acute hepatitis, such as abdominal pain, nausea and vomiting, jaundice, dark urine, and/or light stools within 90 days prior to study entry.
* Peripheral neuropathy greater than or equal to Grade 2 within 90 days prior to study entry according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
* Current cardiovascular disorder that is clinically relevant in the opinion of the site investigator, including but not limited to heart failure, coronary heart disease, second or third degree atrioventricular (AV) block, prolongation of the QRS complex over 120 ms (in both male and female participants), arrhythmia, or tachyarrhythmia.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment including parenteral therapy (e.g., antibiotics) and/or hospitalization within 30 days prior to study entry.
* Currently receiving other medication with potential for adverse drug-drug interactions, including QT prolongation. Please see the study protocol for a list of prohibited medications.
* Taken an investigational drug or vaccine within 30 days prior to study entry.
* Has a clinical condition that in the site investigator's opinion would interfere with study participation.
* Has enrolled into a TB vaccine or TB preventive therapy or TB therapeutic trial, including the A5300B/I2003B/PHOENIx trial, in the two years prior to study entry.
* Not expected to be able to complete 96 weeks of study follow-up (e.g., seasonal or migrant workers or students who may not stay in the area).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5832 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with confirmed or probable active TB at any time between Day 0 and the week 96 study visit | Measured through Week 96
  TB diagnoses will be reviewed by the independent outcomes review committee to assess whether the HHC had TB, if it was confirmed or probable TB, and if it was MDR-TB.
Percent of participants who permanently discontinue randomized study drug (DLM or INH) due to a treatment-related adverse event | Measured through Week 96
  Requiring discontinuation as defined in the protocol, or in the opinion of the site investigator is a treatment-limiting adverse event.

SECONDARY OUTCOMES:
Percent of participants with confirmed active MDR-TB at any time between Day 0 and the week 96 study visit | Measured through Week 96
  Percent of participants with confirmed active MDR-TB at any time between Day 0 and the week 96 study visit
Percent of participants who died from any cause at any time between Day 0 and 96 weeks of follow-up | Measured through Week 96
  Deaths will be reviewed by the independent outcomes review committee to assess whether the HHC had TB at the time of death, possibly undiagnosed, and relatedness of the death to TB.
Percent of participants who died from any cause at any time between Day 0 and 96 weeks of follow-up, or with confirmed or probable active TB at any time between Day 0 and the week 96 study visit | Measured through Week 96
  Deaths and TB diagnoses will be reviewed by the independent outcomes review committee to assess whether the HHC had TB at the time of death, possibly undiagnosed, and relatedness of the death to TB; and whether the HHC had TB, if it was confirmed or probable TB, and if it was MDR-TB.
Percent of participants with a Grade 3 or higher adverse event during the period receiving randomized study drug (DLM or INH) | Measured through Week 26
  If a HHC has a Grade 3 or higher adverse event prior to starting randomized study drug, then the same event will only be considered during follow-up if the grade worsens.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Churchyard, MBBCh MMed FRCP FCP(SA) PhD, Study Chair — Aurum Institute; Amita Gupta, MD, MHS, Study Chair — Johns Hopkins Medical Institutions, Center for Clinical Global Health Education; Anneke Hesseling, MD, PhD, Study Chair — University of Stellenbosch; Susan Swindells, MBBS, Study Chair — University of Nebraska
Locations (31):
- Gaborone CRS, Gaborone, South-East District, Botswana
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Haiti (2):
  - GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS, Port-au-Prince
  - Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince
- India (2):
  - Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra
  - YRG CARE CRS [Site ID: 32075], Chennai, Tamil Nadu
- Kenya (2):
  - Moi University Clinical Research Center (MUCRC) CRS, Eldoret, Rift Valley
  - Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS, Kericho, Rift Valley
- Peru (3):
  - Socios En Salud Sucursal Perú CRS, Lima
  - Barranco CRS, Lima
  - San Miguel CRS, Lima
- De La Salle Health Science Institute Angelo King Medical Research Center (DLSHSI-AKMRC), Cavite, Philippines
- South Africa (10):
  - Soweto ACTG CRS, Johannesburg, Gauteng
  - Wits Helen Joseph Hospital CRS (Wits HJH CRS), Johannesburg, Gauteng
  - Durban International Clinical Research Site CRS, Durban, KwaZulu-Natal
  - PHRU Matlosana CRS, Klerksdorp, North West
  - Rustenburg CRS, Rustenburg, North West
  - Desmond Tutu TB Centre - Stellenbosch University (DTTC-SU) CRS, Cape Town, Western Cape
  - Task Applied Science (TASK) CRS, Cape Town, Western Cape
  - University of Cape Town Lung Institute (UCTLI) CRS, Cape Town, Western Cape
  - South African Tuberculosis Vaccine Initiative (SATVI) CRS, Cape Town, Western Cape
  - CAPRISA eThekwini CRS, Durban
- Kilimanjaro Christian Medical Centre (KCMC), Moshi, Tanzania
- Thailand (3):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Pathum Wan, Bangkok
  - Siriraj Hospital ,Mahidol University NICHD CRS, Bangkok, Bangkoknoi
  - Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Mai
- Uganda (2):
  - Joint Clinical Research Centre (JCRC)/Kampala Clinical Research Site, Kampala
  - MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala
- Vietnam (2):
  - National Lung Hospital CRS (Site ID: 32483), Vĩnh Phúc, Hanoi
  - Vietnam-University of Sydney CRS Site# 32495, Hochiminh City
- Milton Park CRS, Milton Park, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.